CLINICAL TRIAL: NCT03441334
Title: High Frequency Repetitive Transcranial Magnetic Stimulation (rTMS) Combined With Body Weight Supported Treadmill Training (BWSTT) After Stroke: A Pilot Study
Brief Title: rTMS Combined With BWSTT in Stroke With Body Weight Supported Treadmill Training (BWSTT) After Stroke
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The enrollment was not achieved within proposed timeframe.
Sponsor: Texas Woman's University (Other)
Responsible Party: Principal Investigator, Hui Ting Goh, Assistant Professor, Texas Woman's University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19883
Record Dates: First submitted 2018-02-09; First posted 2018-02-22 (Actual); Results first posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- High Frequency rTMS (Experimental): The High Frequency rTMS group will receive real repetitive transcranial magnetic stimulation (rTMS) in 5Hz at 90% of resting motor threshold delivered to the bilateral motor areas via a figure of 8 air-filmed coil. The stimulation is structured as 24 10-second trains with a inter-train interval of 30 second.
  Interventions: Device: High Frequency rTMS
- Sham rTMS (Sham Comparator): The Sham rTMS group will receive the same protocol but delivered via a sham coil which generates the same auditory and cutaneous feedback as the real stimulation. However, there will be no active stimulation.
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: High Frequency rTMS — Participants in the intervention group will receive 1200 stimuli at the intensity of 90% of resting motor threshold via an air-filmed coil placed on the vertex. The stimulation will be delivered across 24 sessions (in 10 weeks). Right after each session, participants will receive a 45-minute structured body weight supported treadmill training.
  Arms: High Frequency rTMS
Device: Sham rTMS — Participants in the sham group will receive the same duration of stimulation via a sham coil placed on the vertex.Right after each session, participants will receive a 45-minute structured body weight supported treadmill training.
  Arms: Sham rTMS

SUMMARY:
The study will enroll 5 individuals post-stroke to examine the feasibility and efficacy of a high frequency repetitive transcranial magnetic stimulation (rTMS) combined with body weight supported treadmill training.

DETAILED DESCRIPTION:
The purpose of this pilot study is to examine the feasibility and efficacy of 5Hz repetitive transcranial magnetic stimulation (rTMS) applied to bilateral motor areas as an adjuvant intervention to task-specific body weight supported treadmill training (BWSTT) in individuals with subacute stroke.

Five individuals with a diagnosis of subacute stroke will be recruited and assigned to either high frequency or sham rTMS group.Both groups will receive a comprehensive assessment of their motor function, gait performance and neurophysiological function before the training. Both groups will then go through a 10 week (24 sessions) of gait training with body weight supported treadmill. For the high frequency rTMS group, they will receive 5 Hz rTMS applied to bilateral motor areas prior to each gait training session. For the sham rTMS group, they will receive a sham stimulation prior to the gait training sessions. All participants will receive another comprehensive assessment after the training concludes. The assessor will be blinded to the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years old
2. < 2 months post stroke at the time of enrollment
3. first time stroke:
4. able to walk > 25 feet with or without assistive device and with no more than moderate assistance:
5. able to follow 1-step commands
6. able to communicate verbally

Exclusion Criteria:

1. severe medical problems (e.g. recent cardiac infarct, heart failure, cancer)
2. presence of conditions that could affect gait training (e.g. amputation, severe arthritis)
3. bilateral stroke
4. non-ambulatory prior to stroke
5. BMI > 40
6. any contraindications to TMS (e.g. history of seizure, cardiac pacemaker, metal or magnetic implants)
7. pregnant or potentially to be pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2018-11-26 (Actual); Study Completion 2018-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Ting Goh, Principal Investigator — Texas Woman's University
Locations (1):
- Texas Woman's University, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High Frequency rTMS | Sham rTMS
Started | 1 (Participant was enrolled in November 2018. Intervention started November 13 2018.) | 0 (no participant enrolled for the sham group)
Completed | 0 (Participant did not complete the protocol. The last treatment session was 11/26/2018) | 0
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: No participants were enrolled for the Sham rTMS group
Groups:
- Total: Total of all reporting groups
Arm/Group | High Frequency rTMS | Sham rTMS | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (0) |  | 58 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 0
  Male | 1 |  | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 1 |  | 1
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Walking Speed
Description: Participant's regular and fast walking speeds (in m/s) will be measured using GaitRite. A faster walking speed indicates a better gait performance.
Time Frame: 10 weeks
Population: We only enrolled 1 participant and the participant did not finish the protocol. We only collected baseline data but not post-training data. The changes in outcome could not be calculated.
Arm/Group | High Frequency rTMS | Sham rTMS
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Quality of Life
Description: Quality of life will be measure using Stroke Impact Scale (SIS). The SIS is a paper and pencil questionnaire consisting 59 items grouped into 8 domains. Each item is rated on a 5-point Likert scale; a higher item score indicates a lower level of difficulty experienced with the item. Item scores are averaged and transformed into domain scores ranging from 0 to 100. A higher domain score indicates a lower level of difficulty. The SIS is well-validated in stroke.
Time Frame: 10 weeks
Population: as for outcome 1
Arm/Group | High Frequency rTMS | Sham rTMS
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Motor Function
Description: Motor function will be quantified using Fugl-Meyer Motor Assessment. The Fugl-Meyer Assessment is well-validated in stroke and has a total score ranging from 0 to 100. A higher total score suggests a better level of motor function.
Time Frame: 10 weeks
Population: as for outcome 1
Arm/Group | High Frequency rTMS | Sham rTMS
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Cortical Excitability
Description: Cortical excitability will be measured using single pulse transcranial magnetic stimulation. Excitability will be quantified using motor evoked potential amplitude (in mV). A higher motor evoked potential amplitude indicates a greater level of excitability.
Time Frame: 10 weeks
Population: as for outcome 1
Arm/Group | High Frequency rTMS | Sham rTMS
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Walking Endurance
Description: Walking endurance will be measured using Six Minute Walk Test and measured in meters. A higher score in the 6 minute walk test (in meters) indicates a better walking endurance.
Time Frame: 10 weeks
Population: as for outcome 1
Arm/Group | High Frequency rTMS | Sham rTMS
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 weeks The only enrolled participant started on November 12 2018 and withdrew on November 26 2018. Participant was monitored via emails and texts up to 2 weeks after the last session (Nov 26 2018)
Arm/Group | High Frequency rTMS | Sham rTMS
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-04): https://cdn.clinicaltrials.gov/large-docs/34/NCT03441334/Prot_SAP_004.pdf